CLINICAL TRIAL: NCT01958385
Title: A RANDOMIZED, SUBJECT AND EVALUATOR-BLINDED, PARALLEL-GROUP, MULTICENTER CLINICAL TRIAL USING AN ENDOSCOPIC SUTURING DEVICE (G-CATH EZ™ SUTURE ANCHOR DELIVERY CATHETER) FOR PRIMARY WEIGHT LOSS
Brief Title: The USGI Medical ESSENTIAL Study for Weight Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: USGI Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G130163
Record Dates: First submitted 2013-10-04; First posted 2013-10-09 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Obesity
Keywords: Total Body Weight Loss
MeSH Terms: conditions — Obesity | interventions — Diet; Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Treatment group (Active Comparator): The treatment of obese patients with the placement of g-Cath EZ suture anchors along with Diet and Exercise
  Interventions: Device: placement of g-Cath EZ suture anchors; Behavioral: Diet and Exercise
- Sham Group (Sham Comparator): The treatment of obese patients with the sham procedure along with Diet and Exercise
  Interventions: Procedure: Sham procedure; Behavioral: Diet and Exercise

INTERVENTIONS:
Device: placement of g-Cath EZ suture anchors
  Other Names: g-Cath EZ™ Suture Anchor Delivery Catheter (USGI Medical)
  Arms: Treatment group
Procedure: Sham procedure
  Arms: Sham Group
Behavioral: Diet and Exercise — A structured diet and exercise plan

SUMMARY:
This is a multicenter, randomized, evaluator and subject blinded, parallel-group, controlled study intended to evaluate the safety and efficacy of treating obese patients with the placement of g-Cath EZ suture anchors followed by a structured diet and exercise plan as compared to a sham procedure followed by the same diet and exercise plan. Subjects will be randomly assigned in a 2:1 ratio to the treatment procedure followed by diet and exercise or the sham procedure followed by diet and exercise. After un-blinding at 12 months post-treatment, sham patients can choose to have the treatment procedure as well.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent.
2. Be male or female subjects between the ages of 22-60 years.
3. If female, be either post-menopausal, surgically sterile or agree to practice birth control during year of study and have negative serum HCG at screening and baseline.
4. Have a Body Mass Index (BMI) of ≥30 and <35 with at least one non-severe co-morbid obesity related condition or a BMI ≥ 35 and < 40 with or without a non-severe obesity related co-morbid condition, where a severe co-morbid condition is defined as severe if symptoms cause severe discomfort, performance of daily activities is compromised, and/or condition is not entirely controlled with prescription drug therapy.
5. Have had no significant weight change (+/- 5% of total body weight) in last 6 months.
6. Have an American Society Anesthesiologists-PS score ≤ 2 (Appendix III).
7. Agrees not to have any additional weight loss interventional procedures, liposuction, or take any over the counter or prescription weight loss medication for 24 months following study enrollment.
8. Have not taken any prescription or over the counter weight loss medications for at least 6 months and agrees not to utilize for 12 months following study enrollment.
9. Be willing to cooperate with post-operative dietary recommendations and assessment tests.
10. Reside within a reasonable distance from the Investigator's treating office (~50 miles) and able and willing to travel to the Investigator's office to complete all routine follow-up visits.

Exclusion Criteria:

1. History of (or intra-operative evidence of) prior bariatric, gastric or esophageal surgery.
2. Esophageal stricture or other anatomy and/or condition that could preclude passage of endolumenal instruments.
3. Severe gastro-esophageal reflux disease (GERD), defined as symptoms that cause subject severe discomfort, compromise performance of daily activities, and/or condition is not entirely controlled with prescription drug therapy.
4. Large hiatal hernia (>3 cm) by history or as determined by pre-randomization endoscopy.
5. Pancreatic insufficiency/disease.
6. Active gastric erosions or gastric/duodenal ulcer.
7. History of gastroparesis or symptoms that would be suggestive of gastroparesis.
8. Pregnancy or plans of pregnancy in the next 12 months.
9. Immunosuppressive medications or systemic steroids (i.e., oral prednisone) within 1 month of Visit 1. Intranasal/inhaled steroids are acceptable.
10. History of inflammatory disease of the GI tract; coagulation disorders; hepatic insufficiency or cirrhosis
11. History or present use of insulin or insulin derivatives for treatment of diabetes
12. Type II Diabetes Mellitus (as defined by HgbA1c >6.5%) for greater than 10 years at the time of enrollment
13. Quit smoking within the last 6 months at time of enrollment or plans to quit smoking in the year after enrollment
14. Portal hypertension and/or varices.
15. Gastric outlet obstruction or stenosis.
16. Significant abnormality identified during Visit 2 (randomization visit) with endoscopy revealing large hiatal hernia, gastric ulcer, gastric erosions, etc.
17. Patient has a history of drug or alcohol abuse or positive at screening for drugs of abuse.
18. Beck Depression Inventory (Short) Score ≥12 and/or uncontrolled depression after pre-enrollment psychological and medical assessment.
19. Present or past history of psychosis, bipolar disease, or obsessive compulsive disorder after pre-enrollment history and medical /psychological assessment.
20. Non-ambulatory or has significant impairment of mobility.
21. Known hormonal or genetic cause for obesity with the exception of treated hypothyroidism.
22. Participating in another clinical study.
23. Is a relative of investigator or his/her staff, or is employed by investigator or institution involved in the study.
24. Subjects with a personal history of allergic/anaphylactic reactions including hypersensitivity to the drugs or materials that will be utilized in the study procedure.

Ages: 22 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 377 (Actual)
Dates: Start 2013-12-01 (Actual); Primary Completion 2015-05-01 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Total Body Weight Loss | Enrollment to 12 months
  Evaluate the effectiveness of the g-Cath EZ™ Suture Anchor Delivery Catheter (USGI Medical, San Clemente, CA, USA) with diet and exercise as an early weight loss intervention for Class I obesity subjects with at least one non-severe obesity related co-morbid condition or Class II obesity subjects with or without a non-severe obesity related co-morbid condition compared to a sham procedure, diet and exercise group.

SECONDARY OUTCOMES:
Quality of Life scores (IWQOL) | enrollment to 12 months
  Assessment of changes
Comorbid status | Enrollment to 12 months
  Assessment of changes from baseline at 12 months in hypertension, diabetes, and hyperlipidemia
Eating Behavior changes | Enrollment to 12 months
  assessment of changes from baseline at 12 months in eating behavior scores (TFEQ) and subjective changes in food capacity, hunger, and satiety in both study groups

CONTACTS AND LOCATIONS:
Overall Officials: Tom Lavin, MD, Principal Investigator — Crescent City Surgical Center
Locations (11):
- United States (11):
  - Scottsdale Healthcare, Scottsdale, Arizona
  - DeWitt Daughtry Family Department of Surgery University of Miami Miller School of Medicine, Miami, Florida
  - Hamilton Medical Center, Dalton, Georgia
  - NorthShore University HealthSystem, Evanston, Illinois
  - Crescent City Surgical Centre, Covington, Louisiana
  - Brigham & Women's Hospital, Boston, Massachusetts
  - University of MN, Fairview Health Services, Minneapolis, Minnesota
  - Saint Luke's Hospital, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Lexington Medical Center, West Columbia, South Carolina
  - Baptist Memorial, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sullivan S, Swain JM, Woodman G, Antonetti M, De La Cruz-Munoz N, Jonnalagadda SS, Ujiki M, Ikramuddin S, Ponce J, Ryou M, Reynoso J, Chhabra R, Sorenson GB, Clarkston WK, Edmundowicz SA, Eagon JC, Mullady DK, Leslie D, Lavin TE, Thompson CC. Randomized sham-controlled trial evaluating efficacy and safety of endoscopic gastric plication for primary obesity: The ESSENTIAL trial. Obesity (Silver Spring). 2017 Feb;25(2):294-301. doi: 10.1002/oby.21702. Epub 2016 Dec 21. PMID 28000425